CLINICAL TRIAL: NCT06140082
Title: Study on the Association of GSTP1 and Other Gene Polymorphisms With Platinum-induced Myelosuppression
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: LI YAN (Other)
Responsible Party: Sponsor-Investigator, LI YAN, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: QFS-LY-2022-GSTP1-001
Record Dates: First submitted 2023-10-04; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gene mutation-type group: According to the characteristics of the patient's own disease, the clinician develops the corresponding medication regimen, and the patient uses one of the target drugs, cisplatin/carboplatin/nedaplatin/loplatin, or other regimen containing the target drug. Peripheral blood of patients was collected, genetic testing was performed, GSTP1 mutant (AG/GG) was classified into this group, and the time and degree of myelosuppression in this group were recorded.
- Gene wild-type group: According to the characteristics of the patient's own disease, the clinician develops the corresponding medication regimen, and the patient uses one of the target drugs, cisplatin/carboplatin/nedaplatin/loplatin, or other regimen containing the target drug. Peripheral blood of patients was collected for genetic testing, GSTP1 wild type (AA) was classified into this group, and the time and degree of myelosuppression in this group were recorded.
  Interventions: Genetic: GSTP1 A313G （AA）

INTERVENTIONS:
Genetic: GSTP1 A313G （AA） — Patients with pulmonary malignant tumors receiving platinum-containing chemotherapy regimen were included in the retrospective and prospective bidirectional cohort study to collect the basic information of the subjects, including gender, age, smoking history, primary site, basic liver and kidney function, chemotherapy regimen, etc. The polymorphisms of glutathione S transferase (GSTP1 A313G) were detected by Sanger dideoxy termination sequencing. The wild type (AA) and mutant type (AG/GG) were divided into two groups.
  Groups: Gene wild-type group

SUMMARY:
This study intends to design a retrospective and prospective, cohort study to explore the association between genetic polymorphism of GSTP1 A313G rs1695 or others and adverse effects of platinum drugs, aiming to explore the risk factors of myelosuppression caused by platinum drugs, and provide data support for optimizing anti-tumor chemotherapy regimen, improve medication safety and improve the compliance of chemotherapy in patients.

DETAILED DESCRIPTION:
Patients with pulmonary malignant tumors receiving platinum-containing chemotherapy regimen were included in the retrospective and prospective bidirectional cohort study to collect the basic information of the subjects, including gender, age, smoking history, primary site, basic liver and kidney function, chemotherapy regimen, etc. The polymorphisms of glutathione S transferase (GSTP1 A313G) were detected by Sanger dideoxy termination sequencing. To study the risk factors related to myelosuppression during chemotherapy, and to preliminarily explore the characteristics of myelosuppression caused by combination chemotherapy with platinum.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with non-small cell lung cancer with clear imaging or pathological evidence
2. Using a chemotherapy regimen containing platinum
3. Conducted blood routine and biochemical tests
4. Signed informed consent

Exclusion Criteria:

1. Blood routine and other relevant tests were not performed
2. Suffering from primary bone marrow system disease
3. Other reasons for not meeting the experimental requirements

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with non-small cell lung cancer with clear imaging or pathological evidence are treated with a platinum-containing chemotherapy regimen
Sampling Method: Non-Probability Sample
Enrollment: 477 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of myelosuppression (≤150 days) | The platinum-based regimen was followed by 4 to 6 cycles of chemotherapy (each cycle is 28 days), 4 visits per treatment cycle, and day0, day1, day2-5, day6-21 after chemotherapy were recorded
  Myelosuppression was judged according to WHO grading criteria

CONTACTS AND LOCATIONS:
Overall Officials: Peng Jing, doctor, Principal Investigator — Jining Medical University; Guo Nan, doctor, Principal Investigator — Shandong Provincial Hospital; Guo LuBo, doctor, Principal Investigator — Jinan Municipal Central Hospital; Liu Lun, doctor, Principal Investigator — Tai 'an City Central Hospital; Zhang ZongLin, doctor, Principal Investigator — Linyi People's Hospital; Di HuiFeng, doctor, Principal Investigator — Jinan Municipal People's Hospital; Sun DeQing, doctor, Principal Investigator — The Second Hospital of Shandong University; Zhang XiaoLi, doctor, Principal Investigator — Shandong Province Third hospital; Liu JianFang, doctor, Principal Investigator — People's Hosital of Rizao; si JiGang, doctor, Principal Investigator — Zibo Central Hospital; Chen HaiSheng, doctor, Principal Investigator — Shandong Provincial Tumor Hospital; Bi HengTai, doctor, Principal Investigator — Weifang Central Hospital